CLINICAL TRIAL: NCT02641977
Title: Longterm Followup of Patients With Rheumatoid Arthritis Treated With Methotrexate Enroled in the Ratingener Rheuma-Kohorte
Brief Title: Longterm Followup of Patients With Rheumatoid Arthritis Treated With Methotrexate
Acronym: MTX
Status: Completed | Type: Observational
Sponsor: Ruhr University of Bochum (Other)
Responsible Party: Principal Investigator, Dietmar Krause, MD, Principal investigator, Ruhr University of Bochum
Other Study IDs: 19802015
Record Dates: First submitted 2015-12-06; First posted 2015-12-30 (Estimated); Last update posted 2018-10-19 (Actual); Status verified 2018-10

CONDITIONS: External Causes of Morbidity and Mortality

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Longterm followup of patients with rheumatoid arthritis 30 years after starting a baseline treatment with Methotrexate.

DETAILED DESCRIPTION:
Objective. 30-year follow-up of rheumatoid arthritis (RA) patients treated with methotrexate (MTX) in the 1980s to analyze the association of the degree of response to MTX with long-term mortality.

Methods. In this observational cohort study, 271 RA patients who had started treatment with MTX between 1980 and 1987 were included (mean age 58 years, mean disease duration 8.5 years). One year after baseline, the treatment response to MTX was evaluated. Responders were defined as patients with at least 20% improvement. Thereafter, assessments were performed at 10 and 18 years after baseline. This re-evaluation was done to provide the data after 30 years of follow-up. Standardized mortality ratios (SMR) are calculated, Cox regression and logistic regression are performed.

ELIGIBILITY:
Inclusion Criteria:

* rheumatoid arthritis
* treatment with methotrexate
* active disease

Exclusion Criteria:

* low disease activity
* previous treatment with methotrexate

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: patients with rheumatoid arthritis
Sampling Method: Non-Probability Sample
Enrollment: 271 (Actual)
Dates: Start 2015-08; Primary Completion 2016-04 (Actual); Study Completion 2016-08 (Actual)

PRIMARY OUTCOMES:
mortality | 30 years

CONTACTS AND LOCATIONS:
Overall Officials: Dietmar MJ Krause, MD, Principal Investigator — University Bochum, Germany
Locations (1):
- Internistische und rheumatologische Praxis Gladbeck, Gladbeck, Germany

IPD SHARING:
Plan to Share IPD: No